CLINICAL TRIAL: NCT01181219
Title: Behandling av Keratoconus Med "Cornea Collagen Cross-linking" Uten Hornhinneepitelfjerning
Brief Title: Transepithelial Corneal Collagen Cross-linking (CXL) in Treatment of Keratoconus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXL-TE UNN2010
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2012-05

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CXL without epithelial removal (Experimental): Application of Riboflavin and the consequent UV-irradiation with intact corneal epithelium
  Interventions: Procedure: CXL without epithelial removal
- CXL with epithelial removal (Active Comparator): Corneal epithelial removal prior to Riboflavin and the consequent UV-irradiation
  Interventions: Procedure: CXL with epithelial removal

INTERVENTIONS:
Procedure: CXL without epithelial removal — UV-radiation of a Riboflavin saturated cornea without prior epithelial removal
  Arms: CXL without epithelial removal
Procedure: CXL with epithelial removal — UV-radiation of a Riboflavin saturated cornea after surgical epithelial removal has been performed
  Arms: CXL with epithelial removal

SUMMARY:
Transepithelial CXL (performed without epithelial removal) seem to have similar clinical effect on keratoconic eyes compared to the standard CXL (which includes epithelial removal). The current study attempts to prove that hypothesis.

A prospective, controlled, randomized, contralateral trial, will involve one eye of the patient to be treated with transepithelial CXL, while the control eye will be treated with the standard CXL. Totally 20 patients (age >18 and <40 years) referred by an ophthalmologist to the eye department of the University Hospital North Norway for CXL treatment of bilateral progressive keratoconus, will be recruited.

DETAILED DESCRIPTION:
CXL appears to hinder the development of keratoconus by strengthening the cross-bindings in the corneal stroma with a resultant increase in corneal biomechanical strength of up to 300%. The method was introduced in the mid-nineties and has been approved for use in the EU countries since 2007. Standard treatment protocol, involving the removal of the corneal epithelium before the Riboflavin application, has been used. In order to avoid potential complications following removal of the epithelium (infection, delayed healing, scar formation, as well as discomfort and pain), a modified procedure where the epithelium is kept intact, so called transepithelial CXL, has been suggested. According to the preliminary results of the published retrospective studies, no significant difference in the clinical effect between the standard CXL with epithelial removal and the transepithelial CXL was found.

ELIGIBILITY:
Inclusion Criteria:

* Documented keratoconus progression in both eyes during the last 12 months before the treatment - decrease in best spectacle-corrected visual acuity (BSCVA) and/or increase in cornea curvature or asymmetry
* Corneal thickness ≥400μm at the thinnest point
* Age range from 18 to 40
* Amsler-Krumeich classification graded stage I to III

Exclusion Criteria:

* Corneal thickness <400μm at the thinnest point
* History of viral keratitis
* Severe dry eye
* Concurrent corneal infections
* Previous ocular surgery
* Hard contact lens wear for ≤4 weeks before baseline examination

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Best corrected distant visual acuity (BCDVA) | One year

SECONDARY OUTCOMES:
Corneal topographic keratoconus features | One year
  Corneal topographic features (and indices) showing keratectatic development will be followed (K-values, optical asymmetry, posterior surface protrusion and thickness).

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Stojanovic, MD, Principal Investigator — University Hospital North Norway
Locations (1):
- University Hospital North Norway, Tromsø, Troms, Norway

REFERENCES:
- [Derived] Stojanovic A, Zhou W, Utheim TP. Corneal collagen cross-linking with and without epithelial removal: a contralateral study with 0.5% hypotonic riboflavin solution. Biomed Res Int. 2014;2014:619398. doi: 10.1155/2014/619398. Epub 2014 Jun 22. PMID 25050368